CLINICAL TRIAL: NCT04515589
Title: Central Aspects of Pain in Rheumatoid Arthritis
Acronym: CAP-RA
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Versus Arthritis (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20001
Record Dates: First submitted 2020-08-06; First posted 2020-08-17 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Pain; Fatigue; Central Sensitization
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main study cohort: The main study cohort in this single-arm cohort is 250 adults with rheumatoid arthritis

SUMMARY:
This study seeks to measure the psychometric properties of a newly developed Central Aspects of Pain in Rheumatoid Arthritis (CAP-RA) questionnaire, and investigate the ability of this questionnaire to measure central mechanisms of pain and also to predict worse pain and fatigue outcomes in people with Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
Persistent pain and fatigue are prevalent and disabling symptoms in people with Rheumatoid Arthritis, even in the absence of active inflammation. The investigators believe that these symptoms may be a result of abnormal pain processing by the Central Nervous System (CNS), in a process called central sensitization.

The investigators have developed a short, self-report questionnaire to measure central pain mechanisms in people with RA. It is called Central Aspects of Pain in Rheumatoid Arthritis (CAP-RA), and was adapted from a pre-existing questionnaire called CAP-Knee (which measures central sensitization in people with chronic knee pain).

This study aims to measure the psychometric properties of CAP-RA, and the ability of the questionnaire to predict worse pain in the RA population. Secondary objectives of the study include predicting worse fatigue in people with RA, deriving CAP-RA scoring recommendations, investigating other factors associated with persistent RA pain, the association between central sensitization and pain, and investigating the course of pain and fatigue in RA.

Participants will be recruited from a Rheumatology clinic. At baseline and 12 weeks these participants will undergo quantitative sensory testing (QST, pain tests), ultrasound for synovitis, clinical assessments, laboratory tests for systemic inflammation and, complete a questionnaire booklet, including the CAP-RA questionnaire.

Some participants will complete the CAP-RA questionnaire 1 week after the baseline visit to assess the test-retest reliability of the questionnaire.

In addition, participants will provide weekly pain and fatigue self-report via text message (SMS) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age≥18y) of any sex and ethnicity.
* Satisfy EULAR criteria for RA.
* Active RA, as defined as DAS28 ≥3.2 at baseline visit

Exclusion Criteria:

* Unable to give informed consent.
* Insufficient understanding of spoken or written English to comply with the requirements of the study protocol
* Unable or unlikely to complete the proposed 12-week study follow up (eg. moving house, terminal diagnosis, current or planned pregnancy).
* Active comorbidity (e.g. uncontrolled diabetes mellitus, cancer, infection) requiring changes in medical treatment at baseline
* Major active psychiatric condition (e.g. major depression)
* Inability to meet the requirements of clinical assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include people with Rheumatoid Arthritis receiving care at the Kings Mill Hospital, Sherwood Forest NHS Foundation Trust, Nottinghamshire, UK, who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Psychometric properties of CAP-RA | Baseline
  A detailed assessment of the psychometric properties of CAP-RA. Higher scores indicate stronger central mechanisms of pain.
Psychometric properties of CAP-RA | 1 week test-retest
  A detailed assessment of the psychometric properties of CAP-RA. Higher scores indicate stronger central mechanisms of pain
Bodily pain | 12 weeks
  Numerical Rating Scale (0-10) of bodily pain - increasing severity

SECONDARY OUTCOMES:
Quantitative Sensory Testing | Baseline
  Validation of CAP-RA as a measure of central sensitization. Lower pressure pain detection thresholds indicate greater sensitivity to painful stimulation. Higher temporal summation indicates dysfunctional pain response. Higher conditioned pain modulation indicates more dysfunctional pain response.
Quantitative Sensory Testing | 12 weeks
  Validation of CAP-RA as a measure of central sensitization. Lower pressure pain detection thresholds indicate greater sensitivity to painful stimulation. Higher temporal summation indicates dysfunctional pain response. Higher conditioned pain modulation indicates more dysfunctional pain response.
Fatigue | 12 weeks
  Bristol Rheumatoid Arthritis Multidimensional Fatigue Scale (BRAFS). 0-70 scale of increasing fatigue.
Change and trajectory of bodily pain | 12 weeks
  Responses to mobile phone text messages giving 0-10 pain scores.
Change and trajectory of fatigue | 12 weeks
  Responses to mobile phone text messages giving 0-10 fatigue scores
Physical activity | 12 weeks
  International Physical Activity Questionnaire (IPAQ) -short form. Lower scores indicate less physical activity.
Functional status | 12 weeks
  Health Assessment Questionnaire (HAQ). Range 0-3 with higher scores indicating greater disability.
Neuropathic pain mechanisms | 12 weeks
  PainDETECT. Higher scores indicating greater neuropathic pain mechanisms.
Mental health | 12 weeks
  Hospital Anxiety and Depression Scale (HADS) - depression and anxiety. Higher scores indicating worse feelings of anxiety and lower mood.
Central sensitization | 12 weeks
  Central Sensitisation Inventory 9 (CSI-9). Higher scores indicate greater central sensitisation.
Joint inflammation | 12 weeks
  Ultrasound assessment showing synovitis
Swollen joints | 12 weeks
  Swollen joint count (0-28)
Inflammation-Erythrocyte sedimentation rate | 12 weeks
  Erythrocyte sedimentation rate (mm per hour)
Inflammation-CRP | 12 weeks
  High sensitivity C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: David A Walsh, Principal Investigator — University of Nottingham
Locations (1):
- Sherwood Forest Hospitals NHS Foundation Trust, Mansfield, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pre-planned analyses will be performed by the study team. Requests for collaborative analyses of IPD, using non-identifiable data, may be made to the study PI.

REFERENCES:
- [Derived] Ifesemen OS, McWilliams DF, Ferguson E, Wakefield R, Akin-Akinyosoye K, Wilson D, Platts D, Ledbury S, Walsh DA. Central Aspects of Pain in Rheumatoid Arthritis (CAP-RA): protocol for a prospective observational study. BMC Rheumatol. 2021 Jun 24;5(1):23. doi: 10.1186/s41927-021-00187-2. PMID 34162435